CLINICAL TRIAL: NCT02168361
Title: The SIM-SOF Trial: A Randomized Trial Comparing Simeprevir-Sofosbuvir Versus Peginterferon/Ribavirin/Sofosbuvir for the Treatment of Chronic Hepatitis C Genotype-1a-infected Patients With Cirrhosis
Brief Title: The SIM-SOF Trial for Hepatitis C
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Center For Hepatitis C, Atlanta, GA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHC-21
Record Dates: First submitted 2014-06-17; First posted 2014-06-20 (Estimated); Results first posted 2016-03-04 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Chronic Hepatitis C
Keywords: cirrhosis
MeSH Terms: conditions — Hepatitis C, Chronic; Fibrosis | interventions — peginterferon alfa-2b; Simeprevir; Ribavirin; Sofosbuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard (Active Comparator): Pegylated Interferon Alfa-2b (1.5 ugm/kg/week subcutaneously) plus ribavirin (1000-1200 mg daily orally) plus sofosbuvir (400 mg daily) for 12 weeks
  Interventions: Drug: Pegylated Interferon alfa-2b; Drug: Ribavirin; Drug: Sofosbuvir
- Simeprevir + Sofosbuvir (Experimental): (SIM-SOF) which is Simeprevir + Sofosbuvir for 12 weeks
  Interventions: Drug: Simeprevir; Drug: Sofosbuvir

INTERVENTIONS:
Drug: Pegylated Interferon alfa-2b — 1.5 ugm/kg/week subcutaneously injected along with ribavirin and sofosbuvir for 12 weeks total
  Other Names: Pegintron
  Arms: Standard
Drug: Simeprevir — 150 mg daily orally along with pegylated interferon and sofosbuvir for a total of 12 weeks
  Other Names: Olysio
  Arms: Simeprevir + Sofosbuvir
Drug: Ribavirin — 1000-1200 mg daily divided twice daily for 12 weeks in combination with pegylated interferon and sofosbuvir
  Other Names: Ribavirin Ribasphere Ribapak
  Arms: Standard
Drug: Sofosbuvir — 12 weeks of combination sofosbuvir and simeprevir
  Other Names: Sovaldi

SUMMARY:
Randomized trial of Hepatitis C-genotype 1-infected patients with compensated cirrhosis comparing the standard of care (Peginterferon/Ribavirin/Sofosbuvir) versus the off-label combination of simeprevir+ sofosbuvir without Ribavirin.

DETAILED DESCRIPTION:
Patients can be treatment naive or prior null response to Peg/RBV, and must be genotype subtype 1a.

Must have Child's Class A cirrhosis/compensated and no history of decompensation

ELIGIBILITY:
Inclusion Criteria:

* chronic hepatitis c,
* cirrhosis biopsy-proven, or via fibrotest,
* CPT score less than 7,
* genotype 1a,
* INR 2.3 or less,
* serum albumin greater than 2.7 gm/dL,
* total bilirubin less than 3 gm/dL,
* platelet count 50,000 per cubic milliliter or more
* GFR >50 ml/min

Exclusion Criteria:

* non genotype 1a,
* history of CPT class B or C or decompensation or history of same,
* HIV or HBV coinfection,
* prior treatment with boceprevir, telaprevir or any other direct acting antiviral agent,
* uncontrolled psychiatric or cardiopulmonary disorders,
* planning pregnancy or unwilling/unable to practice contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2013-12; Primary Completion 2014-12 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian L Pearlman, MD, Principal Investigator — Center for Hepatitis C
Locations (1):
- Center for Hepatitis C, Atlanta, Georgia, United States

REFERENCES:
- [Result] Pearlman BL, Ehleben C, Perrys M. The combination of simeprevir and sofosbuvir is more effective than that of peginterferon, ribavirin, and sofosbuvir for patients with hepatitis C-related Child's class A cirrhosis. Gastroenterology. 2015 Apr;148(4):762-70.e2; quiz e11-2. doi: 10.1053/j.gastro.2014.12.027. Epub 2014 Dec 31. PMID 25557952

RESULTS

PARTICIPANT FLOW:
Groups:
- All Oral Therapy: Simeprevir-sofosbuvir
- Interferon-containing Arm: Peginterferon/ribavirin/sofosbuvir
Period: Overall Study
Arm/Group | All Oral Therapy | Interferon-containing Arm
Started | 62 | 31
Completed | 57 | 21
Not Completed | 5 | 10

BASELINE CHARACTERISTICS:
Population: All participants that received at least a single dose of medication
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Therapy Arm | Interferon-containing Arm | Total
Number analyzed (Participants) | 58 | 24 | 82
Age, Customized [Number; unit: participants]
  Younger than 18 years old | 0 | 0 | 0
  18 years or older | 58 | 24 | 82
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 9 | 29
  Male | 38 | 15 | 53

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Sustained Virologic Response 12 (SVR-12)
Description: Undetectable virus (sensitive nucleic acid test) in Serum at 3 months post-therapy
Time Frame: 12 weeks post-therapy
Population: All participants that received at least a single dose of medication
Measure: Number; unit: participants
Arm/Group | All Oral Therapy | Interferon-containing Arm
Number analyzed (Participants) | 58 | 24
participants | 54 | 18
Statistical Analysis 1: Comparison: All Oral Therapy vs Interferon-containing Arm; Null hypothesis is no difference between two regimens in SVR-12; Test type: Superiority or Other; p = .02, Chi-squared

2. Secondary Outcome: Serum HCV RNA Level
Time Frame: 4 and 12 weeks into therapy
Population: All participants that received at least a single dose of medication
Measure: Median (Full Range); unit: IU/ml
Arm/Group | All Oral Therapy | Interferon-containing Arm
Number analyzed (Participants) | 58 | 24
IU/ml
  Serum HCV RNA level at 4 weeks | 154 [0 to 3000] | 880 [0 to 8500]
  Serum HCV RNA level at 8 weeks | 31 [0 to 112] | 740 [0 to 6050]

ADVERSE EVENTS:
Arm/Group | All Oral | Interferon-containing
Serious Adverse Events (participants affected / at risk) | 0/58 | 1/24
Other Adverse Events (participants affected / at risk) | 46/58 | 22/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Oral (N=58) | Interferon-containing (N=24)
liver decompensation (Hepatobiliary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Oral (N=58) | Interferon-containing (N=24)
rash (Skin and subcutaneous tissue disorders) | 10 | 3
pruritus (Skin and subcutaneous tissue disorders) | 6 | 4
insomnia (Nervous system disorders) | 3 | 6
nausea (Gastrointestinal disorders) | 6 | 7
fatigue (General disorders) | 8 | 17
headache (Nervous system disorders) | 7 | 8
asthenia (Gastrointestinal disorders) | 0 | 4
back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
fever (General disorders) | 0 | 5
flu like illness (General disorders) | 0 | 6
myalgia (Musculoskeletal and connective tissue disorders) | 2 | 4
diarrhea (Gastrointestinal disorders) | 1 | 2
irritability (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
neutropenia (500-750/mm3) (Blood and lymphatic system disorders) | 0 | 4
anemia (Blood and lymphatic system disorders) | 1 | 9
thrombocytopenia (Blood and lymphatic system disorders) | 0 | 3
high bilirubin (Hepatobiliary disorders) | 4 | 0
high amylase (Gastrointestinal disorders) | 12 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No